CLINICAL TRIAL: NCT06159816
Title: PREVALENCE STUDY OF PNH CLONES IN PATIENTS WITH NEOPLASIES MYELOPROLIFERATIVE PHILADELPHIA-NEGATIVE
Brief Title: PREVALENCE STUDY OF PNH CLONES IN PATIENTS WITH NEOPLASIES
Status: Completed | Type: Observational
Sponsor: AUSL Romagna Rimini (Other)
Responsible Party: Sponsor
Other Study IDs: MyeloPNH
Record Dates: First submitted 2023-11-20; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Myeloproliferative Neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicenter prevalence study of the PNH clone (paroxysmal hemoglobinuria nocturnal) in SMP Ph-. This multicenter, prospective study aims to evaluate the presence of an PNH clone in patients with a confirmed diagnosis of myeloproliferative neoplasia Phcon or without mutations in the 3 main genes involved in this disease (JAK2, MPL, and Cal-R),but showing signs of ongoing hemolysis or particular clinical conditions.

To this end, a multicolor flow cytometric test will be used to evaluate the presence of deficient GPI molecules in granulocytic, monocytic and other cells erythrocyte (flow cytometric test, based on the use of the FLAER reagent in peripheral blood samples).

The study will be conducted at clinical hematology centers in the wider area of the Romagna and at other Italian hematology clinical centers, where and analyzed the peripheral blood samples and clinical data to be included in the study.

The participating centers will carry out the flow cytometric diagnostic test at i own reference laboratories, while the biological material for subsequent studies genetic-molecular type (next generation sequencing) will be analyzed centrally at the Biosciences laboratory of the IRST IRCCS only for cases testing positive for the presence of the PNH clone. Clinical information will be collected for each patient enrolled in the study necessary for the classification of the case and all the laboratory data necessary for achievement of the objectives of the study. The main objective of the study is to evaluate the prevalence of PNH clones in patients with a confirmed diagnosis of myeloproliferative neoplasm Ph- with or without mutations affecting the 3 main genes involved in this disease (JAK2, MPL, e Cal-R), but showing signs of ongoing hemolysis or particular clinical conditions.

Secondary objectives of the study are:

- correlate the characteristics of the PNH clone with the clinical characteristics and laboratory of myeloproliferative neoplasms Ph- (the presence of phenomena thrombotics, the disease state, the DIPSS prognostic score index, and the state mutational).

· characterize the genomic architecture of the cases using NGS technology positive results

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of one of the following Ph-negative myeloproliferative neoplasms:

   polycythemia vera, essential thrombocythemia, idiopathic myelofibrosis, according to i WHO 2016 criteria
2. Women or men, age ≥ 18 years.
3. Willingness and ability to give written informed consent and adhere to study procedures.
4. Availability of the result of the following molecular tests:

   * JAK2-V617F mutation,
   * JAK2 exon 12 in PV (if JAK2 negative) Cal-R, and MPL in MFI and TE (if JAK2 negative)
5. Obvious signs of hemolysis (defined as LDH≥1.5 x ULN, reduced haptoglobin, reticulocytosis) when not related to the underlying disease or significantly changed compared to baseline values OR Detection of a thrombotic event (subsequent to diagnosis) OR Appearance or worsening of anemia OR Symptom change (appearance or worsening of signs or symptoms) in a stable disease context.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of one of the following Ph-negative myeloproliferative neoplasms:
  polycythemia vera, essential thrombocythemia, idiopathic myelofibrosis, according to i WHO 2016 criteria
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
the prevalence of PNH clones | 2022
  evaluate the prevalence of PNH clones in patients with a confirmed diagnosis of myeloproliferative neoplasm Ph- with or without mutations affecting the 3 main genes involved in this disease (JAK2, MPL, e Cal-R), but showing signs of ongoing hemolysis or particular clinical conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Ausl Della Romagna, Ravenna, Italy

REFERENCES:
- [Derived] D'Addio A, Rondoni M, Salvucci M, Marconi G, Bonifacio M, Tanasi I, Perbellini O, Carli G, Tosi P, Tomassetti S, Poletti G, Massari E, Rosetti M, Fabbri E, Zingaretti C, Lucchesi A, Bochicchio MT, Simonetti G, Krampera M, Lanza F. PNH clones prevalence study in ph-negative myeloproliferative neoplasms: a multicenter Italian study. Ann Hematol. 2025 Sep;104(9):4487-4494. doi: 10.1007/s00277-025-06556-y. Epub 2025 Aug 22. PMID 40844514